CLINICAL TRIAL: NCT07064616
Title: Pulsed Field Ablation vs. Cryoballoon Ablation in Patients With Persistent Atrial Fibrillation
Acronym: PEACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kitasato University (Other)
Collaborators: Nerima Hikarigaoka Hospital (Unknown); Sagamihara Kyodo Hospital (Unknown)
Responsible Party: Principal Investigator, Hidehira Fukaya, Junior Associate Professor, Kitasato University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C24-157
Record Dates: First submitted 2025-07-05; First posted 2025-07-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-06

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Pulsed-field ablation; Cryoballoon ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed-Filed Ablation (PFA) group (Active Comparator): The PFA group includes persistent AF patients treated with PFA
  Interventions: Device: Catheter ablation using pulsed field ablation
- Cryoballoon (CBA) group (Active Comparator): The CBA group includes persistent AF patients treated with CBA
  Interventions: Device: Catheter ablation using cryoballoon ablation

INTERVENTIONS:
Device: Catheter ablation using pulsed field ablation — PulseSelect™ Pulsed Field Ablation System:
  This intervention uses the PulseSelect™ system to perform pulsed field ablation (PFA) for pulmonary vein isolation in patients with persistent atrial fibrillation. PFA delivers short, high-voltage electrical pulses that selectively affect myocardial cells while minimizing damage to surrounding tissues such as the esophagus or phrenic nerve. This technique is designed to reduce procedural complications and improve safety compared to traditional thermal ablation methods.
  Arms: Pulsed-Filed Ablation (PFA) group
Device: Catheter ablation using cryoballoon ablation — Cryoballoon Ablation:
  This intervention uses a cryoballoon catheter to perform pulmonary vein isolation by freezing tissue around the pulmonary veins. The balloon delivers extreme cold temperatures to create transmural lesions that block abnormal electrical signals responsible for atrial fibrillation. Cryoballoon ablation is widely used and considered effective for atrial fibrillation treatment but may carry risks related to collateral tissue injury.
  Arms: Cryoballoon (CBA) group

SUMMARY:
This clinical study is being conducted to compare two different treatment methods for persistent atrial fibrillation (AF), a common heart rhythm disorder. Atrial fibrillation occurs when the upper chambers of the heart (the atria) beat rapidly and irregularly. This can lead to symptoms like palpitations, shortness of breath, or fatigue, and it increases the risk of stroke or heart failure.

Persistent atrial fibrillation means that the irregular heart rhythm continues and does not stop on its own. Treatment often includes a procedure called catheter ablation, where special instruments are used to create small scars in the heart to block the abnormal electrical signals causing the arrhythmia.

Currently, two main types of catheter ablation are used in Japan:

Cryoballoon Ablation: A technique that uses extreme cold to create scars and isolate the pulmonary veins, which are often the source of the irregular signals.

Pulsed Field Ablation (PFA): A newer technique that uses very short bursts of electrical energy to target the heart tissue, with the aim of reducing damage to surrounding structures.

While pulsed field ablation has been introduced in Japan recently and seems to be safe, there is limited data about how well it works compared to cryoballoon ablation, especially in patients with persistent atrial fibrillation. This study aims to find out whether pulsed field ablation is as effective and safe as cryoballoon ablation for treating persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Diagnosed with PeAF (lasting less than one year or requiring cardioversion)
* Eligible for catheter ablation according to current Japanese guidelines
* Provided written informed consent

Exclusion Criteria:

* Paroxysmal or long-standing persistent AF (duration >1 year)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation recurrence at 12 months | 12 months post-procedure
  Proportion of patients without documented atrial fibrillation lasting 30 seconds or longer after a 3-month blanking period following the ablation procedure, assessed by ECG or Holter monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Kitasato University School of Medicine, Sagamihara, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: Undecided